CLINICAL TRIAL: NCT07349446
Title: Effects of Circadian-Based Acupressure on Sleep Quality in Nursing Home Residents: A Randomized Controlled Trial
Brief Title: Effects of Circadian-Based Acupressure on Sleep Quality in Nursing Home Residents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Krida Wacana Christian University (Other)
Responsible Party: Principal Investigator, Santa Maria Pangaribuan, Principal Investigator, Registered Nurse, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 001/KEPK/IKI/E2/I/2026; NSTC113-2628-B-038-003-MY3 (Other Grant/Funding Number: Taiwan's National Science and Technology Council); NSTC114-2314-B-038-094-MY3 (Other Grant/Funding Number: Taiwan's National Science and Technology Council); 01/UKKW/LPPM-FKIK/LIT/I/2026 (Other Grant/Funding Number: Universitas Kristen Krida Wacana)
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Poor Sleep Quality; Anxiety; Depression; Stress; Insomnia
Keywords: poor sleep quality; Insomnia; depression; anxiety; stress
MeSH Terms: conditions — Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Two arm parallel group designs: (1) Circadian-based acupressure intervention, and (2) Sham acupressure.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant will be blinded to group allocation. Outcome assessors will remain blinded to group allocation until the end of the study, therapists will be aware of group assignments due to the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circadian-based acupressure (Experimental): Participants in the Circadian-based Acupressure group will receive circadian-based acupressure twice daily, five days a week for four weeks.
  Interventions: Other: Circadian-based acupressure
- Sham Acupressure (Sham Comparator): Sham Acupressure (placebo) group received massage at a non-acupuncture point.
  Interventions: Other: Sham Acupressure

INTERVENTIONS:
Other: Circadian-based acupressure — Participants in the Circadian-based Acupressure group will receive circadian-based acupressure twice daily, five days a week for four weeks. Acupressure will be administered in the morning one hour after breakfast (at 11am) and in the evening one to two hours before bedtime (at 7 pm). Acupressure was performed by applying consistent fingertip pressure of 3-5 kg, with gentle rotational movements, on the selected acupoints. The selected acupoints were based on our network meta-analysis the most used acupoint: Sanyinjiao (SP6), Shenmen (HT7), Fengchi (GB20), and Neiguan (PC6). The accuracy of the acupressure was confirmed if the participants felt sore, numb, distended, or warm at the point of application. The duration of each session was limited to 3 minutes, with an interval of 5 seconds of pressure followed by a 1-second rest. Acupoints of Sanyinjiao and Shenmen will be apply at 11 am and Neiguan and Fengchi at 7 pm.
  Arms: Circadian-based acupressure
Other: Sham Acupressure — Sham Acupressure (placebo) group received massage at a non-acupuncture point, located 10 mm from the actual point, with the same frequency as the experimental group. According to traditional Chinese medicine, manipulation of non-acupuncture points should not elicit a sensation of de qi.
  Arms: Sham Acupressure

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of circadian-based acupressure compared with sham acupressure in improving sleep quality among nursing home residents. Additionally, the study will examine the effects of the intervention on insomnia severity, heart rate variability, and psychological distress, including depression, anxiety, and stress. A total of 80 older adults aged 60 years and above residing in a nursing home in Jakarta, Indonesia, will be randomly assigned to either the circadian-based acupressure group or the sham acupressure group. Participants in the intervention group will receive circadian-based acupressure twice daily, five days per week for four weeks, with acupoints selected and administered according to circadian meridian activity, while the control group will receive sham acupressure at non-acupuncture points with the same frequency and duration. Outcome measures will be assessed at baseline and immediately post-intervention.

DETAILED DESCRIPTION:
Poor sleep quality affects approximately 65% of institutionalized older adults and is associated with adverse outcomes including cognitive decline, psychological distress, falls, and increased mortality. Current geriatric guidelines recommend nonpharmacological interventions as first-line management for sleep disturbances. Acupressure, a low-cost and non-invasive therapy derived from Traditional Chinese Medicine (TCM), has shown promise in improving sleep; however, prior trials have largely used fixed protocols without considering circadian timing. According to TCM meridian clock theory, qi circulates through specific meridians in a 24-hour rhythm, suggesting that time-aligned acupressure may enhance therapeutic effects. To evaluate the effectiveness of circadian-based acupressure on sleep quality in nursing home residents compared with sham acupressure, and to examine its effects on insomnia severity, heart rate variability (HRV), depression, anxiety, and stress. This randomized, participant- and assessor-blinded controlled trial will recruit 80 nursing home residents aged ≥60 years in Jakarta, Indonesia. Eligible participants must have lived in the facility for ≥3 months, score ≥25 on the Mini-Mental State Examination, and have poor sleep quality (PSQI ≥5). Participants will be randomly assigned (1:1) to circadian-based acupressure or sham acupressure. The intervention will be delivered twice daily, five days per week for four weeks: SP6 and HT7 at 11:00 am, and PC6 and GB20 at 7:00 pm, aligning with circadian meridian activity. Each acupoint will be stimulated for 3 minutes using standardized pressure. The sham group will receive massage at non-acupoints with identical frequency and duration. The primary outcome is sleep quality measured by the Pittsburgh Sleep Quality Index (PSQI). Secondary outcomes include insomnia severity (Athens Insomnia Scale), HRV (ANSWatch), and psychological distress (DASS-21). Measurements will be collected at baseline and immediately post-intervention (Week 4). Analyses will follow the intention-to-treat principle. Baseline differences will be assessed using chi-square tests, ANOVA, or nonparametric equivalents. Intervention effects over time will be examined using generalized estimating equations to assess group × time interactions, adjusting for demographic covariates. Post-hoc pairwise comparisons will be conducted when appropriate. Missing data will be handled using multiple imputation. Statistical significance will be set at p ≤ 0.05. This study is the first randomized controlled trial to investigate circadian-based acupressure in nursing home residents. Findings will provide evidence on whether aligning acupressure with circadian meridian activity enhances sleep quality and related physiological and psychological outcomes, supporting a feasible and theory-driven nonpharmacological intervention for institutionalized older adults.

ELIGIBILITY:
Inclusion Criteria:

* age ≥60 years
* ability to communicate and complete the questionnaires in Indonesian
* had lived in the nursing home for at least 3 months,
* had a Mini-Mental State Examination score of ≥25, had self-reported PSQI Indonesian version scores of ≥5 (where higher scores indicate worse sleep) over the past 4 weeks,
* agreed to participate in the research

Exclusion Criteria:

* The exclusion criteria in this study were severe psychiatric disorders, such as schizophrenia, bipolar disorder, or current receipt of intensive psychiatric treatment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | Baseline (before intervention/0 weeks) and After Intervention (4 weeks)
  Sleep quality was measured using the Pittsburgh Sleep Quality Index (PSQI). The PSQI can be used to assess self- reported sleep quality and sleep disturbance in the preceding month. The scale comprises 19 items and the following seven dimensions: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) sleep efficiency, (5) sleep disturbance, (6) sleeping medication use, and (7) daytime dysfunction. The items are rated on a four-point Likert scale with endpoints ranging from 0 to 3, and the overall score ranges from 0 to 20. A score of less than five indicates favorable sleep quality. The Indonesian version of the PSQI exhibited high validity and reliability (Cronbach's α = 0.720)

SECONDARY OUTCOMES:
Insomnia | Baseline (before intervention/0 weeks) and After Intervention (4 weeks)
  Insomnia was measured using Athens Insomnia Scale. The AIS-8 is an eight-item self-report questionnaire that measures the intensity of sleep difficulties (Soldatos et al., 2000, 2003) in accordance with the ICD-10 diagnostic criteria for insomnia. Five items assess sleep induction, awakenings during the night, final awakening earlier than desired, total sleep duration, and overall sleep quality. Total scores for the AIS-8 range from 0 to 24. The AIS Indonesian demonstrated favorable internal consistency (Cronbach's α: 0.86), and acceptable test-retest reliability (0.85). CFA indicated a strong model fit for the AIS-I. AIS-I scores exhibited significant associations with the ISCI, IGAD-7, and IPHQ-9, and EQ-5D (r = -0.55, 0.55, 0.66, and -0.31, respectively, all P < .001). Scores greater than 7 were classified as indicating insomnia.
Heart Rate Variability | Baseline (before intervention/0 weeks) and After Intervention (4 weeks)
  HRV was measured using a wrist monitor ANSWatch model (TS-0411, Taiwan Scientific Corp., Taipei, Taiwan). ANSWatch was calibrated using a sphygmomanometer U-300 with an accuracy of ±8 mmHg, and calibrated using ECG (Agilent A3) with an accuracy of ±5%
Psychological distress | Baseline (before intervention/0 weeks) and After Intervention (4 weeks)
  Psychological distress was measured using the Depression, Anxiety and Stress Scale (DASS-21) Bahasa Indonesia version. It is translated by Damanik (2011). This is a self-report questionnaire consists of three 14-items subscales, measure depression, anxiety and stress (negative mental health). Total score ranged from 0-42 with higher scores showing higher level of distress.

CONTACTS AND LOCATIONS:
Overall Officials: Santa Maria Pangaribuan, M.Sc, Principal Investigator — Taipei Medical University, Taiwan
Locations (1):
- Jl. Bina Marga No.58 7 6 7, RT.7/RW.5, Cipayung, Kec. Cipayung, Kota Jakarta Timur, Daerah Khusus Ibukota Jakarta 13840, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Particular data will be shared: Individual participant data that underlie the results reported in this article after identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 60 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose, for example, for a meta-analysis or other study.

REFERENCES:
- [Background] Soldatos CR, Dikeos DG, Paparrigopoulos TJ. The diagnostic validity of the Athens Insomnia Scale. J Psychosom Res. 2003 Sep;55(3):263-7. doi: 10.1016/s0022-3999(02)00604-9. PMID 12932801
- [Background] Soldatos CR, Dikeos DG, Paparrigopoulos TJ. Athens Insomnia Scale: validation of an instrument based on ICD-10 criteria. J Psychosom Res. 2000 Jun;48(6):555-60. doi: 10.1016/s0022-3999(00)00095-7. PMID 11033374
- [Background] Setyowati A, Chung MH. Validity and reliability of the Indonesian version of the Pittsburgh Sleep Quality Index in adolescents. Int J Nurs Pract. 2021 Oct;27(5):e12856. doi: 10.1111/ijn.12856. Epub 2020 Jul 7. PMID 32632973
- [Background] Schlaeger JM, Gabzdyl EM, Bussell JL, Takakura N, Yajima H, Takayama M, Wilkie DJ. Acupuncture and Acupressure in Labor. J Midwifery Womens Health. 2017 Jan;62(1):12-28. doi: 10.1111/jmwh.12545. Epub 2016 Dec 21. PMID 28002621
- [Background] Reza H, Kian N, Pouresmail Z, Masood K, Sadat Seyed Bagher M, Cheraghi MA. The effect of acupressure on quality of sleep in Iranian elderly nursing home residents. Complement Ther Clin Pract. 2010 May;16(2):81-5. doi: 10.1016/j.ctcp.2009.07.003. Epub 2009 Aug 19. PMID 20347838
- [Background] Raana HN, Fan XN. The effect of acupressure on pain reduction during first stage of labour: A systematic review and meta-analysis. Complement Ther Clin Pract. 2020 May;39:101126. doi: 10.1016/j.ctcp.2020.101126. Epub 2020 Feb 29. PMID 32379664
- [Background] Geng SH, Liu L, Lin ZM, Zhang H, Mei RG, Liu X, Liu JC, Huang GR, Zhang WC. A review of novel research technology to explore the mystery of traditional Chinese medicine: Terahertz. Medicine (Baltimore). 2023 Nov 17;102(46):e35870. doi: 10.1097/MD.0000000000035870. PMID 37986326
- [Background] Pangaribuan SM, Wu TY, Herlianita R, Jao YL, Lee HC, Hasan F, Mukminin MA, Chiu HY. Global occurrence rates of sleep disturbances among institutionalized older adults: A systematic review and meta-analysis. Sleep Med Rev. 2025 Jun;81:102091. doi: 10.1016/j.smrv.2025.102091. Epub 2025 Apr 11. PMID 40239318
- [Background] Luo J, Feng L, Wang L, Fang Z, Lang J, Lang B. Restoring brain health: Electroacupuncture at GB20 and LR3 for migraine mitigation through mitochondrial restoration. Brain Circ. 2024 Jun 26;10(2):154-161. doi: 10.4103/bc.bc_95_23. eCollection 2024 Apr-Jun. PMID 39036293
- [Background] Li LW, Harris RE, Tsodikov A, Struble L, Murphy SL. Self-Acupressure for Older Adults With Symptomatic Knee Osteoarthritis: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2018 Feb;70(2):221-229. doi: 10.1002/acr.23262. Epub 2017 Dec 29. PMID 28437570
- [Background] Lee WJ, Park H. Effects of auricular acupressure on sleep and pain in elderly people who have osteoarthritis and live in nursing homes: A randomized, single-blind, placebo-controlled trial. Explore (NY). 2023 Mar-Apr;19(2):214-222. doi: 10.1016/j.explore.2022.07.001. Epub 2022 Jul 5. PMID 35835645
- [Background] Lee IS, Ryu Y, Chae Y. Oversimplifying the name of the 12 meridian channels. Integr Med Res. 2023 Dec;12(4):101002. doi: 10.1016/j.imr.2023.101002. Epub 2023 Oct 21. No abstract available. PMID 37953755
- [Background] Lai FC, Chen IH, Chen PJ, Chen IJ, Chien HW, Yuan CF. Acupressure, Sleep, and Quality of Life in Institutionalized Older Adults: A Randomized Controlled Trial. J Am Geriatr Soc. 2017 May;65(5):e103-e108. doi: 10.1111/jgs.14729. Epub 2017 Feb 2. PMID 28152177
- [Background] Hmwe NT, Subramanian P, Tan LP, Chong WK. The effects of acupressure on depression, anxiety and stress in patients with hemodialysis: a randomized controlled trial. Int J Nurs Stud. 2015 Feb;52(2):509-18. doi: 10.1016/j.ijnurstu.2014.11.002. Epub 2014 Nov 11. PMID 25468282
- [Background] Hmwe NTT, Browne G, Mollart L, Allanson V, Chan SW. Acupressure to improve sleep quality of older people in residential aged care: a randomised controlled trial protocol. Trials. 2020 Apr 25;21(1):360. doi: 10.1186/s13063-020-04286-2. PMID 32334620
- [Background] Bourgeois J, Elseviers MM, Van Bortel L, Petrovic M, Vander Stichele RH. Sleep quality of benzodiazepine users in nursing homes: a comparative study with nonusers. Sleep Med. 2013 Jul;14(7):614-21. doi: 10.1016/j.sleep.2013.03.012. Epub 2013 May 18. PMID 23692988